CLINICAL TRIAL: NCT02689726
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, and Immunogenicity of GTL001 Vaccine Adjuvanted With Imiquimod Cream in HPV 16- and/or HPV 18-Infected Women Aged 25 to 65 Years, With Normal Cytology, ASCUS, or LSIL
Brief Title: Safety, Tolerability, and Immunogenicity of GTL001 Vaccine Adjuvanted With Imiquimod Cream in HPV 16- and/or HPV 18-Infected Women Aged 25 to 65 Years, With Normal Cytology, ASCUS, or LSIL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy in European Phase 2 study
Sponsor: Genticel (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC10VAC05; 016462 (Registry Identifier: Serial No.: 0001)
Record Dates: First submitted 2015-06-29; First posted 2016-02-24 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: HPV 16- and/or HPV 18-Infected Women With Normal Cytology, ASCUS, or LSIL
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GTL001 + Aldara, 5% imiquimod cream (Experimental): 2 doses, 6 weeks apart, GTL001 will be adjuvanted with Aldara, 5% imiquimod cream, applied to the injection site 15 minutes and 24 hours after each vaccination
  Interventions: Drug: GTL001+; Drug: Aldara

INTERVENTIONS:
Drug: GTL001+
Drug: Aldara — 5% imiquimod cream

SUMMARY:
A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, and Immunogenicity of GTL001 Vaccine Adjuvanted With Imiquimod Cream in HPV 16- and/or HPV 18-Infected Women Aged 25 to 65 Years, With Normal Cytology, ASCUS, or LSIL.

DETAILED DESCRIPTION:
This is an outpatient, open-label study. After a screening period of up to 4 weeks, all eligible subjects will receive 2 doses, 6 weeks apart, of GTL001 Powder reconstituted with water for injection. GTL001 will be adjuvanted with Aldara, 5% imiquimod cream, applied to the injection site 15 minutes and 24 hours after each vaccination. The follow-up period is 12 weeks from the first injection. The duration of the study is defined for each subject as the date that signed, written informed consent is provided through the last follow-up visit. Total duration of subject participation is approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Females between the ages of 25 and 65 years, inclusive, at the time of screening.
2. Subject is in generally good health based on medical history and on clinically acceptable results, in the judgment of the investigator, on the following assessments: physical examination, vital signs, clinical chemistry, and hematology.
3. Cervical HPV 16 and/or 18 infection confirmed by cobas® HPV Test (Roche Molecular Systems, Inc) real-time polymerase chain reaction (RT PCR) assay at screening.
4. Cervical cytological evaluation with a normal, ASCUS, or LSIL result.
5. Subjects of childbearing potential must use effective contraception at the time of GTL001 injection and for at least 12 months after the first vaccination. Effective methods of birth control include those that result in a low failure rate (ie, less than 1% per year) when used consistently and correctly, such as implants, injectable, combined oral contraceptives, desogestrel only pill, levonorgestrel-releasing intrauterine system, intrauterine devices, vasectomized partner, and true sexual abstinence. Subjects not of childbearing potential include those who are surgically sterile or postmenopausal (no menses for the previous 12 months).
6. Subject is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.
7. In the opinion of the investigator, the subject is able to comply with the protocol and has a high probability of completing the study.

Exclusion Criteria:

1. Current or history of untreated high-grade cervical lesion (either CIN2 or CIN3).
2. Current or history of cervical, vulvar, or vaginal cancer.
3. Prior exposure to HPV prophylactic vaccine, regardless of number of doses received, or participation in another HPV vaccination clinical trial.
4. Current acute or chronic disease, other than HPV 16/18 infection, which would be expected to interfere with the protocol-defined evaluations.
5. Clinically significant gynecological abnormalities that could interfere with study procedures (eg, prolapse, severe vaginal atrophy, myoma, hysterectomy) in the judgment of the investigator.
6. Malignancy, or treatment for malignancy, within the previous 2 years, with the exception of basal cell or squamous cell carcinoma of the skin.
7. Clinically important abnormalities in the physical examination or laboratory tests during the screening period (ie, hemoglobin level <9.5 g/dL, white blood cells <2500 cells/mm3, aspartate aminotransferase and/or alanine aminotransferase ≥1.5 × the upper limit of normal [ULN], creatinine ≥1.25 × ULN, alkaline phosphatase ≥2 × ULN, and total bilirubin >ULN).
8. Administration of any live viral vaccine within 3 months or any inactivated (nonlive) vaccine within 2 weeks prior to screening.
9. Primary or secondary systemic immunosuppression (defined as prolonged [≥7 days] use of corticosteroids that is ≥20 mg/day of prednisone equivalent or any other immunosuppressive drug).
10. History of severe allergy requiring hospital care or history of severe asthma requiring oral or parenteral drug management in the last year.
11. Known hypersensitivity to imiquimod.
12. History of a severe reaction to any drug or vaccination.
13. Medical condition with clinical and/or biological consequences judged by the investigator to be incompatible with ID vaccination.
14. History of, or positive test results at screening for, human immunodeficiency virus, hepatitis B virus surface Ag, or hepatitis C virus.
15. Current episode of symptomatic vaginal or genital infection.
16. Current episode or history of genital herpes.
17. Subject is pregnant or lactating/breastfeeding.
18. Use of any investigational drug within 30 days before screening or current participation in another clinical trial.
19. History of recent (within 1 year) alcohol/drug abuse.
20. Employee or family member of the investigator or study site personnel.
21. Enrollment goals have been reached in the subject's age cohort

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic reactions recorded on diary cards as a measure of safety and tolerability | 14-day period following an injection
  To assess the tolerability, with respect to vaccine-specific local and systemic reactions, of GTL001 adjuvanted with imiquimod in women in 2 age cohorts: 25 to 50 years, inclusive, and 51 to 65 years, inclusive. The diary cards will include local abd systemic reactions to the adjuvant, medications taken with start and stop dates, and other unsolicited symptoms/complaints, including start and stop dates.

SECONDARY OUTCOMES:
Level of anti-CyaA serum as a measure of cellular and humoral Immunogenicity | 12 weeks
  Measured by enzyme-linked immunoabsorbent assay (ELISA) at weeks 0,2,6,8, and 12 (Visits 1,2,3,4, and 5, respectively) To assess the cellular and humoral immunogenicity of GTL001 adjuvanted with imiquimod in the 2 age cohorts.
Percentage of subjects with anti-CyaA serum antibody response as a measure of cellular and humoral immunogenicity | 12 weeks
  Measured at weeks 2,6,8, and 12 (Visits 2,3,4, and 5, respectively) To assess the cellular and humoral immunogenicity of GTL001 adjuvanted with imiquimod in the 2 age cohorts.
Specific responses to HPV 16 and HPV 18 E7 Ag stimulation as a measure of cellular and humoral Immunogenicity | 12 weeks
  Measured at weeks 0,2,6,8, and 12 (Visits 1,2,3,4, and 5, respectively) To assess the cellular and humoral immunogenicity of GTL001 adjuvanted with imiquimod in the 2 age cohorts.
Percentage of subjects with positive specific response to HPV 16 and/or HPV 18 E7 stimulation as a measure of cellular and humoral Immunogenicity | 12 weeks
  To assess the cellular and humoral immunogenicity of GTL001 adjuvanted with imiquimod in the 2 age cohorts.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Louisville, Louisville, Kentucky
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Clinical Research Advantage, Inc./ Columbus Obstetricians and Gynecology, Inc., Columbus, Ohio
  - Planned Parenthood Southeastern Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No